CLINICAL TRIAL: NCT04643652
Title: Effective Strategies to Reduce Noise and Noise Related Distractions in the ICU : a Stepped Wedge Cluster Randomized Controlled Trial
Brief Title: Effective Strategies to Reduce Noise and Related Distractions
Acronym: NOISY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-5541
Record Dates: First submitted 2020-09-08; First posted 2020-11-25 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Noise Exposure; Intensive Care Unit; Safety Issues
Keywords: Noise; ICU; Alarms; Annoyance; Distractions

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Cluster Randomised Model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual Care
- Intervention (Experimental): Implementation of a Noise Reduction Bundle
  Interventions: Behavioral: Noise Reduction Bundle

INTERVENTIONS:
Behavioral: Noise Reduction Bundle — Implementation of a bundle of noise reducing interventions. This concerns among other things:
  reduction of alarms, phone calls/pagers/ beepers, introduction of a defined period in which there is a reduction of controllable sound (quiet time), etc
  Arms: Intervention

SUMMARY:
Patients admitted to the intensive care unit (ICU) undergo complex critical care treatment and are consequently surrounded by equipment and monitors contributing to high sound pressure levels. In addition, many medical and nursing ICU staff members work together with numerous visiting consultants resulting in an additional sound burden. As is already known, in the ICU environment, many activities carried out by healthcare professionals, require a high level of concentration. So, the noisy ICU environment causes interruptions in activities that require concentration and induce in this way, a higher potential for errors. The World Health Organization (WHO) and the Environmental Protection Agency (EPA) set standards for sound levels in hospitals with a recommendation for patient treatment areas. There is a clear trend for increasing hospital noise since the sixties. According to healthcare professionals, one of the strongest contributing factors of noise in the ICU environment are monitoring alarms as they occur very frequently. Additionally, ICU nurses experience high levels of stress towards clinical alarms and are becoming alarm fatigue, which means that the staff becomes desensitized because of an excessive number of alarms and may disable or silence alarms without checking the patient . Consensus dictates the importance of reducing sound pressure levels and the numerous alarm signals from monitor alarms in the ICU. In the study, we focus on busy predetermined areas in the ICU.

This study aims to determine the effect of an intervention bundle, aimed at the reduction of "noise" (decibels) and its effect on health care professionals.

DETAILED DESCRIPTION:
Design:

The introduction is done by a stepped wedge cluster randomized design. The study will be carried out in five units of the department of intensive care medicine of the Radboud University Medical Center, a 950-bed university hospital in the Netherlands. The study focus on health care providers in the ICU.The research consists of the introduction of an intervention bundle to reduce noise and therefore interruptions during their daily work activities.

Inclusion:

All health care providers present at the ICU, during the study period (about 350) are asked to participate. They will receive information about the aim, content and relevance of the study and will be asked for participation.They are free to refuse to participate in the study (e.g. part of observations, survey).

Methods:

The data collection focuses on quantitative noise measurements at the predetermined locations in ICU units during the study period. In addition, during the entire study period (control and intervention), we analyse the amount and type of alarms. Thirdly, we collect data with regard to disruptions during the daily work process of healthcare professionals (e.g. during "high-risk moments", such as: medication preparation) by observations.

Finally, health care providers are asked about their perceived annoyance, as a result of ambient noise (NRS-annoyance).

Data analysis will be supported with the use of Excel, Phyton and SPSS.

ELIGIBILITY:
Inclusion Criteria:

• Healthcare providers present during the study period (about 250) are asked to participate between august 2022 and december 2023.

Exclusion Criteria:

• Healthcare providers who do not speak / read the Dutch language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Sound pressure levels | through study completion, an average of 1 year
  Sound pressure levels at predetermined locations
Acoustic alarms | through study completion, an average of 1 year
  e.g. acoustic alarms (ventilation, heartrate, tension, etc )

SECONDARY OUTCOMES:
Interruptions | through study completion, an average of 1 year
  e.g. number of interruptions during daily work (count)
Annoyance (as an emotional impact on health care providers) | through study completion, an average of 1 year
  e.g. perceived annoyance caused by alarms, telephones, pagers, conversation

CONTACTS AND LOCATIONS:
Overall Officials: Hans vd Hoeven, MD, PhD, Principal Investigator — Radboud UMC, Dep.Intensive Care, Nijmegen, The Netherlands
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No